CLINICAL TRIAL: NCT06885658
Title: Effectiveness of Visual Storytelling Intervention on Antibiotic Adherence in UTI Patients in Pakistan: a Randomized Controlled Trial
Brief Title: Effectiveness of Visual Storytelling Intervention on Antibiotic Adherence in UTI Patients
Acronym: ABR UTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Iltaf Hussain, Principal Investigator, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BZU-FOPDPP-2466
Record Dates: First submitted 2025-02-28; First posted 2025-03-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Uncomplicated Urinary Tract Infection; Patient With Uncomplicated UTI
Keywords: Visual storytelling; Antibiotic Adherence; UTI recurrence

STUDY DESIGN:
Intervention Model Description: This study uses a parallel two-arm randomized controlled trial (RCT) design. Participants will be randomly assigned in a 1:1 ratio to either:
  Intervention group: Receives a visual storytelling intervention designed to improve antibiotic adherence in patients with urinary tract infections (UTIs).
  Control group: Receives standard care, which includes routine verbal or written instructions about antibiotic use.
  The intervention involves the delivery of a sticker affixed on the antibiotic packaging containing visual stories that emphasize the importance of completing the full antibiotic course and the consequences of non-adherence, including antibiotic resistance. The study aims to compare the effectiveness of this intervention with standard care in improving adherence to prescribed antibiotics
Who Masked: Care Provider, Outcomes Assessor
Masking Description: In this study, the participants and site staff delivering the intervention will not be masked, due to the nature of the behavioral intervention (visual storytelling sticker), which participants will be actively engaged with.
  However, the physician who diagnoses the UTI and confirms UTI recurrence will be blinded to the intervention allocation to avoid bias in outcome assessment.
  Additionally, the data analysts (outcome assessor) will be blinded to group assignments. The dataset will be labeled neutrally (e.g., "Group A" and "Group B") to ensure unbiased analysis of the primary and secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Visual Storytelling using stickers (Experimental): In this arm, participants will receive a visual storytelling intervention designed to improve antibiotic adherence. The intervention involves a stickers (affixed to the antibiotic packages) containing simple, visually appealing illustrations that explain how antibiotics work and the consequences of not completing the full course. The story contrasts the positive outcomes of adhering to the treatment with the risks of non-adherence, including the development of antibiotic resistance. Key messages will highlight the importance of completing the prescribed antibiotic course. The intervention is intended to engage patients emotionally and cognitively, enhancing their understanding of antibiotic use and encouraging adherence to the prescribed treatment regimen.
  Interventions: Behavioral: Visual Storytelling Intervention for Antibiotic Adherence
- Control Group: Standard Care for Antibiotic Adherence (No Intervention): The control group will receive the usual standard care for antibiotic adherence, which typically includes verbal or written instructions provided by the healthcare provider about the correct usage of prescribed antibiotics for treating urinary tract infections (UTI). This group will not receive any additional interventions, such as the visual storytelling intervention. The standard care aims to represent the typical approach to UTI treatment, allowing for a comparison of the effectiveness of the visual storytelling intervention against routine practice in improving antibiotic adherence. Participants in this group will also complete the same baseline and follow-up assessments related to knowledge and attitudes about antibiotics and adherence.

INTERVENTIONS:
Behavioral: Visual Storytelling Intervention for Antibiotic Adherence — The intervention involves the use of a visual storytelling approach designed to improve antibiotic adherence in patients diagnosed with urinary tract infections (UTIs). The intervention consists of a sticker featuring simple, visually appealing illustrations and a narrative highlighting the importance of completing the full course of prescribed antibiotics. The story contrasts the positive outcomes of adhering to the treatment with the negative consequences of stopping early, such as increased bacterial resistance. Key messages are reinforced through bold text and visual cues. This intervention aims to engage patients emotionally and cognitively, promoting behavior change by making the concept of antibiotic adherence more relatable and memorable.
  Arms: Intervention Arm: Visual Storytelling using stickers

SUMMARY:
This study aims to evaluate the effectiveness of a visual storytelling intervention in improving antibiotic adherence among adults with urinary tract infections (UTIs). Participants will be randomly assigned to either the intervention group, where they will receive a visual sticker on their antibiotic packaing, explaining the importance of completing their antibiotic course, or the control group, which will receive routine care. The study will measure how well participants follow their prescribed antibiotic regimens and assess their knowledge and attitudes toward antibiotic use. The goal is to determine if visual storytelling can enhance adherence, reduce antibiotic resistance, and improve health outcomes.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will assess the impact of a visual storytelling intervention on antibiotic adherence among adults diagnosed with uncomplicated urinary tract infections (UTIs). The intervention involves a visually engaging sticker that educates patients on the importance of completing their prescribed antibiotic course and the consequences of non-adherence, such as antibiotic resistance. Participants will be randomly assigned to either the intervention or control group, with the control group receiving standard care (e.g., verbal or written instructions). The primary outcome is adherence to the antibiotic regimen, measured by pill counts. Secondary outcomes include UTI recurrence, knowledge about antibiotic use, and attitudes toward antibiotic treatment. Data will be collected at baseline, immediately after the intervention, and at follow-up visits over 1, 3, and 6 months. This study seeks to determine if visual storytelling can improve antibiotic adherence and help combat antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Physician-confirmed diagnosis of uncomplicated urinary tract infection (UTI).
3. Prescribed oral antibiotics (tablet/capsule) for UTI treatment.
4. Willingness to participate in the study and provide informed consent.
5. Ability to complete follow-up assessments and adhere to the study protocol.

Exclusion Criteria:

1. Diagnosed with complicated UTI (e.g., pyelonephritis, sepsis, or structural abnormalities).
2. Multiple comorbidities that require polypharmacy.
3. Cognitive impairment or mental disorders that would interfere with study participation.
4. Pregnant or breastfeeding women.
5. Participation in another clinical trial that could interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Antibiotic adherence | Based on the antibiotic treatment course (3-7 days)
  The primary outcome measure of this study is antibiotic adherence, which will be assessed by tracking the number of prescribed antibiotic pills taken by the participants at the end of their treatment course (typically 3-7 days).
  Adherence will be calculated in two ways:
  Proportional Adherence: The percentage of the prescribed pills that the patient takes will be calculated, expressed as a proportion (number of pills taken/total prescribed).
  Categorical Adherence: Patients will be categorized as "adhered" (if they took ≥90% of the prescribed antibiotics) or "not adhered" (if they took <90% of the prescribed antibiotics).

SECONDARY OUTCOMES:
UTI Recurrence | UTI recurrence will be assessed at 3 months, and 6 months following the initial antibiotic treatment.
  This outcome will assess whether a participant experiences a recurrence of a urinary tract infection (UTI) after completing the prescribed course of antibiotics. Recurrence will be confirmed by a physician based on clinical evaluation and/or laboratory tests. A binary response (Yes/No) will be recorded based on physician confirmation of UTI recurrence.
Knowledge | Knowledge will be assessed at baseline (before the intervention) and at first follow up (3-7 days) 3 months, and 6 months follow-up after the intervention.
  Knowledge Measurement: A 10-item true/false questionnaire will assess the patient's understanding of antibiotic use, antibiotic resistance, and the importance of completing the full antibiotic course. This includes questions like understanding the consequences of not completing antibiotic treatment or misusing antibiotics.
Attitude | Attitude will be assessed at baseline (before the intervention) and at first follow up (3-7 days) 3 months, and 6 months follow-up after the intervention.
  Attitude Measurement: A 5-item Likert scale will assess the patient's attitude towards antibiotics and adherence. Statements such as "Completing the full course of antibiotics is very important" and "I trust the advice given by my doctor regarding antibiotics" will be used to gauge attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Tertiary care hospitals (n = 6), Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Given the sensitive nature of the data, particularly related to participants' health and personal information, ensuring privacy and confidentiality is of paramount importance. Sharing IPD may risk the unintended disclosure of personal identifiers.
  The study has been approved by an institutional ethics board, and the informed consent provided by participants specified the use of their data strictly for the purposes outlined in the study. Sharing IPD outside the approved scope could violate ethical guidelines and regulatory frameworks.

REFERENCES:
- [Derived] Hussain I, Rasool MF, Ullah J, Khan I, Kadirhaz M, Xu M, Tang C, Dong Y, Zhao W, Khan FU, Chang J, Fang Y. Effectiveness of nudge-based visual storytelling in antibiotic adherence in uncomplicated urinary tract infection in Pakistan: protocol for a randomized controlled trial. Trials. 2025 Dec 17. doi: 10.1186/s13063-025-09328-1. Online ahead of print. PMID 41408333